CLINICAL TRIAL: NCT01368601
Title: Effects of Intraoperative Continuous Airway Pressure (CPAP) on the Inflammatory Response of the Lung With Cancer Undergoing Lobectomy. A Randomised Placebo-controlled Trial
Brief Title: Effects of Intraoperative Continuous Airway Pressure (CPAP) on the Inflammatory Response to One-lung Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Lluís Gallart, MD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INFLATOR
Record Dates: First submitted 2011-05-24; First posted 2011-06-08 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; CPAP; PPC; lobectomy; One-lung ventilation
MeSH Terms: conditions — Lung Neoplasms | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (positive airway pressure) (Active Comparator): To evaluate if continuous positive airway pressure(CPAP) on the lung undergoing lobectomy can decrease the inflammatory response PPC (postoperative pulmonary complications).
  Interventions: Procedure: CPAP (Continuous airway pressure)
- Control without CPAP (No Intervention)

INTERVENTIONS:
Procedure: CPAP (Continuous airway pressure) — To evaluate if continuous positive airway pressure (CPAP) on the lung undergoing lobectomy can decrease the inflammatory response and PPC.
  Arms: CPAP (positive airway pressure)

SUMMARY:
This is a randomized placebo-controlled trial studying the effects of intraoperative continuous airway pressure (CPAP) on the inflammatory response of the lung with cancer undergoing lobectomy.

DETAILED DESCRIPTION:
Pulmonary lobectomy induces an inflammatory response of this lung caused by intraoperative atelectasis and re-expansion. This inflammatory response can be attenuated with treatment, also decreasing postoperative pulmonary complications (PPC). Thus, avoiding complete atelectasis with partial insufflation of the lung during surgery could be useful to decrease inflammatory response and PPC.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-80 aged) with American Society of Anesthesiologists physical status I-III, scheduled to undergo elective thoracic surgery with lung resection performed through thoracotomy, and requiring OLV (one lung ventilation)during surgery.

Exclusion Criteria:

* Ongoing treatment with any dose of systemic or topical steroids, acute pulmonary or extrapulmonary infections (elevated C-reactive protein [CRP]), history of recurrent pneumothoraces, previous thoracic surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-05; Primary Completion 2020-06 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Alveolar and plasmatic cytokines measured before and after atelectasis and re-expansion. | From preoperative to postoperative (24h) period.
  Alveolar and plasmatic cytokines measured before and after atelectasis and re-expansion.

SECONDARY OUTCOMES:
Alveolar MICA | From preoperative to postoperative period (24h)
  Alveolar MICA I (major histocompatibility complex (MHC) class I chain related genes) expression measured at the same control times.
CT-Scan | 22-24h after surgery
  Postoperative distribution of well-aerated, non aerated or poorly aerated lung volumes.
Postoperative pulmonary complications (PPC). | Participants will be followed for the duration of hospital stay, an expected average of 10 days.
  PPC.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain